CLINICAL TRIAL: NCT03592407
Title: A Phase 2 Trial of Neoadjuvant Pembrolizumab in Combination With Epacadostat (INCB024360) in Patients With Non-Metastatic Esophageal/Gastroesophageal Squamous Cell and Adenocarcinomas Treated With Neoadjuvant Chemoradiation: A Window-Of-Opportunity Study
Brief Title: Epacadostat and Pembrolizumab Before Surgery in Treating Participants With Stage II-III Esophageal or Gastroesophageal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17302; NCI-2018-00682 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17302 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-04-30; First posted 2018-07-19 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophageal Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (epacadostat, pembrolizumab) (Experimental): Starting 14 days after completion of standard of care chemoradiotherapy, participants receive epacadostat PO BID during weeks 3-8 and pembrolizumab IV over 30 minutes on day 1 of weeks 3 and 6 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Epacadostat; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Pharmacodynamic Study

INTERVENTIONS:
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC

SUMMARY:
This phase II trial studies the side effects of epacadostat and pembrolizumab and to see how well they work before surgery in treating participants with stage II-III esophageal or gastroesophageal cancer. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of the tumor cells to grow and spread. Giving epacadostat and pembrolizumab before surgery may work better in treating participants with stage II-III esophageal or gastroesophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish that the combination of epacadostat and pembrolizumab will lead to an increase in tumor infiltrating cytotoxic T-cells and circulating cytotoxic T cells and a reduction in immunosuppressive Tregs and myeloid-derived suppressor cells (MDSCs) in esophageal/gastroesophageal junction (GEJ) tumors that can arise after treatment with neoadjuvant chemoradiation.

II. To assess safety and tolerability of pembrolizumab and epacadostat (immunotherapy) in this patient population.

SECONDARY OBJECTIVES:

I. To evaluate pathologic complete response rate (path CR) and correlate with tumor T-cell response.

II. To evaluate complete clinical response rate (clinical CR) and subsequent avoidance of esophagectomy and correlate with tumor T-cell response.

III. To evaluate toxicities with the combination of pembrolizumab and epacadostat in this treatment setting.

IV. To evaluate disease-free survival (DFS) and overall survival (OS) in this treatment population.

EXPLORATORY OBJECTIVES:

I. To measure changes in whole genome serum micro ribonucleic acid (miRNA) signatures before and after protocol therapy and correlate with tumor/immune/stromal cell miRNA expression profiling determined by deep sequencing.

II. To assess the role of circulating miR-23a as serum biomarker given its role as an oncomir in esophagastric cancer and reporting in the literature of suppressing tumor cytotoxic T cells in preclinical models.

III. To correlate diversity in the gut microbiome with path CR and clinical CR after treatment with pembrolizumab and epacadostat.

IV. To measure serial plasma kynurenine/tryptophan ratio levels as a pharmacodynamic marker of increased IDO1 activity and response.

V. Association of PD-L1 expression, microsatellite stability and/or IDO1 expression and pathological complete response (pCR) rate.

OUTLINE:

Starting 14 days after completion of standard of care chemoradiotherapy, participants receive epacadostat orally (PO) twice daily (BID) during weeks 3-8 and pembrolizumab intravenously (IV) over 30 minutes on day 1 of weeks 3 and 6 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at one month and then every 3 months in year 1, every 4 months in year 2, and every 6 months in year 3.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted only with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Non-metastatic cancer of the esophagus OR esophagus and gastroesophageal junction (GEJ; tumor extending =< 2 cm into the stomach)
* Confirmed stage II-III diagnosis of one of the following:

  * Squamous cell; OR
  * Adenocarcinoma; OR
  * Mixed adenosquamous carcinoma
* Deemed appropriate for neoadjuvant chemoradiation by the multidisciplinary team (surgeon, medical oncologist, and radiation oncologist)

  * Chemotherapy defined as weekly carboplatin/paclitaxel; AND
  * Radiation defined as external beam radiotherapy defined as: 50.4 gray (Gy) as per institutional and national treatment guidelines
* Deemed appropriate for esophagectomy or repeat endoscopic biopsies if non-operative management is pursued
* Absolute neutrophil count (ANC) >= 1500/mm^3 within 14 days prior to day 1 of study participation/1st endoscopic biopsy
* Platelets >= 100,000/mm^3 within 14 days prior to day 1 of study participation/1st endoscopic biopsy
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN if total bilirubin levels > 1.5 x ULN within 14 days prior to day 1 of study participation/1st endoscopic biopsy
* Aspartate aminotransferase (AST) =< 2 x ULN within 14 days prior to day 1 of study participation/1st endoscopic biopsy
* Alanine aminotransferase (ALT) =< 2 x ULN within 14 days prior to day 1 of study participation/1st endoscopic biopsy
* Creatinine =<1.5 x ULN OR for patients with Creatinine >1.5 x ULN Creatinine clearance of >=60 ml/min per 24 hour urine test or the Cockcroft-Gault formula
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN within 14 days prior to day 1 of study participation/1st endoscopic biopsy
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Female of childbearing potential only: negative urine or serum pregnancy test; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by women of childbearing potential (WOCBP) and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 120 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Immune checkpoint inhibitor(s) (e.g. anti-PD-1, anti-CTLA4)
* Indoleamine-2,3-dioxygenase (IDO) inhibitors
* Radiotherapy within 21 days prior to day 1 of study participation
* Investigational agent within 21 days prior to Day 1 of study participation
* Live-virus vaccination within 30 days prior to Day 1 of study participation
* Systemic cytotoxic chemotherapy, antineoplastic biologic therapy, or major surgery within 21 days of study participation
* Chronic systemic steroid therapy or on any other form of immunosuppressive medication
* Monoamine oxidase inhibitors (MAOI) or any drug associated with MAOI activity
* Any UGT1A9 inhibitors (including acitretin, amitriptyline, androsterone, cyclosporine, dasatinib, diclofenac, diflunisal, efavirenz, erlotinib, estradiol (17-beta), flutamide, gefitinib, gemfibrozil, glycyrrhetinic acid glycyrrhizin, imatinib, imipramine, ketoconazole, linoleic acid supplements, mefenamic acid, and mycophenolic acid, niflumic acid, nilotinib, phenobarbital, phenylbutazone, phenytoin, probenecid)
* Coumarin-based anticoagulants
* Unstable or untreated brain/leptomeningeal metastasis
* Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, or abdominal carcinomatosis (known risks factors for bowel perforation)
* Severe hypersensitivity reaction to treatment with another antibody and/or hypersensitivity to epacadostat excipients
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C (with confirmation of negative hepatitis B surface antigen [HBsAg], hepatitis B virus [HBV] polymerase chain reaction [PCR], and hepatitis C virus [HCV] PCR)
* History of pneumonitis (non-infectious) that required steroids or current pneumonitis
* Known history of active tuberculosis
* Diagnosed with or treated for cancer within the previous two years, other than histologies listed in inclusion criteria or non-melanoma carcinoma of the skin
* Female only: pregnant or breastfeeding
* Any othr condition that would, in the Investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Temporal anti-tumor immune response defined as tumor infiltrating cytotoxic T-cells, circulating T-cells, T regulatory cells (Tregs), and myeloid-derived suppressor cells (MDSCs) in tumor and blood samples | Baseline to 3 years
  Patient demographics and baseline disease/prior treatment characteristics will be summarized using descriptive statistics. Descriptive statistics will be used to summarize the gene expression profile in tissue/blood. Changes in these measures during and after treatment (when measured) will also be summarized by descriptive statistics and tables/plots. Various statistical analyses will be used to explore the association between these gene expression measures (at different time points and the changes over time) with clinical outcomes. For the exploratory correlation of these endpoints with response, analyses comparing groups of participants defined by response may be conducted by two-sample t-test or Wilcoxon rank sum test.
Incidence of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0 | Up to 8 weeks
  All participants evaluable for toxicity will be included in the toxicity analysis. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Pathological complete response (CR) | Up to 3 years
  Will be defined as no residual cancer cells, including lymph nodes under pathologic examination of the surgically resected specimen and/or a Tumor Regression Score of 0 by the College of American Pathologists (CAP) Cancer Protocol for Esophageal Carcinoma. Pathological response will be determined per CAP Cancer Protocols and will utilize a modified Ryan scheme. For pathological CR, all participants evaluable for response will be included in the analysis. Pathological CR rate will be estimated by the proportion of participants achieving pathological CR along with the 95% exact binomial confidence interval.
Clinical complete response | Up to 3 years
  Defined as no radiographic evidence of disease of positron emission tomography/computed tomography (PET/CT) or CT imaging. For clinical CR, all participants evaluable for response will be included in the analysis. Clinical CR rate will be estimated by the proportion of participants achieving clinical CR along with the 95% exact binomial confidence interval.
Incidence of adverse events per CTCAE v 4.0 | Up to 3 years
  All participants evaluable for toxicity will be included in the toxicity analysis. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Disease free survival (DFS) | From start of neoadjuvant therapy up to 3 years
  DFS will be determined using the Kaplan-Meier method.
Overall survival (OS) | From start of neoadjuvant therapy up to 3 years
  OS will be determined using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chao, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California